CLINICAL TRIAL: NCT07141914
Title: A Master Protocol for Semaglutide Effects on Cardiovascular and Obesity-related Outcomes in People With Overweight or Obesity in the Real World
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-8669; U1111-1326-1795 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-08-15; First posted 2025-08-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity; Heart Failure (HF); Atherosclerotic Cardiovascular Disease (ASCVD); Primary Prevention
MeSH Terms: conditions — Overweight; Obesity; Heart Failure; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort: Semaglutide users
  Interventions: Other: No treatment given
- Cohort: Semaglutide Non-users
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given
  Groups: Cohort: Semaglutide users
Other: No treatment given — No treatment given
  Groups: Cohort: Semaglutide Non-users

SUMMARY:
This study aims to evaluate the association of once-weekly semaglutide with the risk of cardiovascular (CV) and other obesity-related clinical outcomes in three study populations (Heart failure (HF), clinical Atherosclerotic Cardiovascular Disease (ASCVD), primary prevention).

This is a retrospective cohort study which includes administrative medical and pharmacy claims linked with clinical and laboratory measurements for participants in the US during January 1, 2016 - December 31, 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with overweight or obesity defined as at least one overweight/obesity indication of a specified body mass index (BMI) more than or equal to (≥) 27.0 kilogram per meter square (kg/m2) and undefined obesity indications, defined by diagnoses and laboratory values, during January 1, 2016 to December 31, 2024
2. Participants with a record indicating the study population of interest during January 1, 2016 to December 31, 2024

1. HF: Diagnosis of HF 2. Clinical ASCVD: Diagnosis or procedure codes indicating:Coronary artery disease (CAD) including acute coronary syndrome (ACS; i.e., myocardial infarction [MI] or unstable angina), stable angina, coronary or other arterial revascularization or intervention, ischemic stroke, transient ischemic attack (TIA), carotid or other arterial stenosis, peripheral arterial disease (PAD) including aortic aneurysm 3. Primary Prevention: Patients at risk for developing ASCVD defined as the presence of more than or equal to (≥) 3 of the following risk factors

1. Smoking history
2. Dyslipidaemia
3. Hypertension
4. Prediabetes
5. Chronic kidney disease (CKD) or evidence of kidney function decline/kidney damage
6. High-sensitivity C-reactive protein (hs-CRP) more than or equal to (≥) 2 milligram per litre (mg/L)

3. Participants who are more than or equal to (≥) 45 years old by December 31, 2024

4. Participants will be divided into the following groups: those who initiate semaglutide on or after the eligibility date and June 4, 2021 (semaglutide users; date of initiation termed the index date) or participants with no evidence of semaglutide usage during January 1, 2016 to December 31, 2024 (non-users; a randomly selected date with ≥ 1 pharmacy claim on or after the eligibility date and June 4, 2021 will be termed the index date)

5. Participant with continuous insurance enrolment eligibility more than or equal to (≥) 12 months prior to the index date (the baseline period)

6. Participants with re-confirmed overweight/obesity indication during the baseline period

Exclusion Criteria:

1. Population specific exclusion criteria:

1. HF and Clinical ASCVD Populations: Diagnosis of end-stage HF
2. Primary Prevention Population: Diagnosis of HF or haemorrhagic stroke, or evidence of clinical ASCVD

2. Participants with a diagnosis of chronic or acute pancreatitis

3. Participants with a diagnosis of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma

4. Participants with end-stage kidney disease (ESKD) including chronic or intermittent haemodialysis or peritoneal dialysis and/or kidney transplant

5. More than or equal to (≥ 2) diagnoses of cancer (excluding non-melanoma skin cancer)

6. Pregnancy in female participants

7. Evidence of diabetes including more than or equal to (≥) 2 diagnoses of type 1 diabetes or more than or equal to (≥) 2 diagnoses of type 2 diabetes on distinct dates, use of a glucose-lowering agent, and/or glycated haemoglobin (HbA1c) laboratory result more than or equal to ≥ 6.5 percent (%)

8. Use of a glucagon-like peptide-1 (GLP-1) or GLP-1/gastric inhibitory polypeptide (GIP) receptor agonist approved for weight management during the baseline period

9. Participants with evidence of bariatric surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to evaluate the association of once-weekly semaglutide with the risk of CV and other obesity-related clinical outcomes in three study populations. This is a retrospective cohort study which includes administrative medical and pharmacy claims linked with clinical and laboratory measurements for participants in the US during January 1, 2016 - December 31, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 285327 (Actual)
Dates: Start 2025-08-29 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Revised 5-Point Major Adverse Cardiovascular Events (MACE-5) (time-to-event) | Index date, earliest of revised MACE-5 and end of follow-up; up to 42 months
  Measured as Months
  Occurrence of any of the following individual component events:
  1. Myocardial infarction (MI)
  2. Stroke
  3. Hospitalization for HF
  4. Coronary revascularization (including coronary artery bypass grafting and percutaneous coronary intervention)
  5. All-cause mortality
  The event date will be the earliest occurrence of one of the individual components.
Revised 3-point Major Adverse Cardiovascular Events MACE-3 (time-to-event) | Index date, earliest of revised MACE-3 and end of follow-up; up to 42 months
  Measured in Months
  Occurrence of any of the following individual component events:
  1. MI
  2. Stroke
  3. All-cause mortality
  The event date will be the earliest occurrence of one of the individual components.

SECONDARY OUTCOMES:
MI (time-to-event) | Index date, earliest of MI and end of follow-up; up to 42 months
  Measured as Months
  A primary diagnosis of MI (identified using International Classification of Disease, 10th Edition, Clinical Modification (ICD-10-CM) diagnosis codes observed during an inpatient (IP) visit).
  The event date will be admission date of the IP visit.
Stroke (time-to-event) | Index date, earliest of stroke and end of follow-up; up to 42 months
  Measured as Months
  A primary diagnosis of stroke, including both ischemic and haemorrhagic, (identified using ICD-10-CM diagnosis codes observed during an IP visit).
  The event date will be the admission date of the IP visit.
Hospitalization for HF (time-to-event) | Index date, earliest of hospitalization for HF and end of follow-up; up to 42 months
  Measured as Months
  A primary diagnosis of HF (identified using ICD-10-CM diagnosis codes observed during an IP visit).
  The event date will be the first observed admission date of the IP visit.
Coronary revascularization (time-to-event) | Index date, earliest of Coronary revascularization and end of follow-up; up to 42 months
  Measured as Months
  Evidence of coronary revascularization in any claim (identified using International Classification of Disease, 10th Edition, Procedure Coding System (ICD-10-PCS), Current Procedural Terminology (CPT), or Healthcare Common Procedure Coding System (HCPCS) procedure codes).
  The event date will be the first observed date of coronary revascularization.
All-cause mortality (time-to-event) | Index date, end of follow-up; up to 42 months
  Measured as Months
  Evidence of death as recorded at the month and year level in Komodo Research Data (KRD) and defined as a death record observed within the last month of follow-up.
  The event date will be the earliest of the end of follow-up (e.g., bariatric surgery within the month of death and last month of follow-up) or the last day of the recorded month of death.
MACE-5 (time-to-event) | Index date, earliest of MACE-5 and end of follow-up; up to 42 months
  Measured as Months
  Occurrence of any of the following individual component events:
  1. MI
  2. Stroke
  3. Hospitalization for HF
  4. Coronary revascularization
  5. CV-related mortality
  The event date will be the earliest occurrence of one of the individual components.
MACE-3 (time-to-event) | Index date, earliest of MACE-3 and end of follow-up; up to 42 months
  Measured as Months
  Occurrence of any of the following individual component events:
  1. MI
  2. Stroke
  3. CV-related mortality
  The event date will be the earliest occurrence of one of the individual components.
CV-related mortality (time-to-event) | Index date, end of follow-up; up to 42 months
  Measured as Months
  Any claim within ≤30 days before the date of death (i.e. the last day of the recorded month of death, where death is observed in the last month of follow- up) of the following operational definition to indicate CV related mortality:
  1. Primary diagnosis of MI
  2. Primary diagnosis of ischemic or haemorrhagic stroke
  3. Primary diagnosis of HF
  4. Evidence of aortic or peripheral arterial revascularization, coronary revascularization, or carotid revascularization or intervention in any claim
  5. Primary diagnosis of CV haemorrhage (excluding haemorrhagic stroke)
  6. Primary diagnosis of other CV conditions including unstable angina, sudden cardiac arrest, cardiogenic shock, & other cerebrovascular & CV events Non-CV-related mortality is defined as all other records of death that are not classified as CV-related mortality.
  The event date will be the earliest of the end of follow-up (e.g. bariatric surgery within the month of death) or the date of death.
Urgent HF visit (time-to-event) | Index date, earliest of urgent HF visit and end of follow-up; up to 42 months
  Measured as Months
  A primary diagnosis of HF (identified using ICD-10-CM diagnosis codes observed during a non-IP visit). Further, at least one the following interventions must be observed in a non-IP claim on the same day as the non-IP visit:
  1. Procedure indicating administration of intravenous diuretics or vasoactive agents (identified using HCPCS procedure codes)
  2. Pharmacy claim for an intravenous diuretic or vasoactive agent (identified using National Drug Codes (NDCs))
  3. Diagnosis of an encounter for mechanical circulatory support or mechanical fluid removal or dependence on dialysis (identified using ICD-10-CM diagnosis codes)
  4. Procedure for mechanical circulatory support or mechanical fluid removal (identified using ICD-10- PCS, CPT, and HCPCS procedure codes)
  The event date will be the first observed date of the non-IP visit that meets the urgent HF criteria.
3-point HF (time-to-event) | Index date, earliest of 3-point HF composite outcome and end of follow-up; up to 42 months
  Measured as Months
  Occurrence of any of the following individual component events:
  1. Hospitalization for HF
  2. Urgent HF visit
  3. CV-related mortality
  The event date will be the earliest occurrence of one of the individual components.
2-point HF (time-to-event) | Index date, earliest of 2-point HF composite outcome and end of follow-up; up to 42 months
  Measured as Months
  Occurrence of any of the following individual component events:
  1. Hospitalization for HF
  2. Urgent HF visit
  The event date will be the earliest occurrence of one of the individual components.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational, Plainsboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com